CLINICAL TRIAL: NCT06867965
Title: A Study to Investigate the Function, Safety and Tolerability of a Subcutaneous Continuous Glucose Monitoring System in Diabetic Patients (Type 1 and 2)
Brief Title: Feasibility Study of a Novel Subcutaneous Continuous Glucose Monitoring System in Diabetics
Acronym: FiberSense
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EyeSense GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: P-4.1-C-0.1
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BellySense system (Experimental): 8 diabetic patients will wear a BellySense system at the upper arm or abdomen for up to 14 days.
  Interventions: Device: BellySense

INTERVENTIONS:
Device: BellySense — BellySense is a novel CGM system, based on a fiber-optical sensor placed through the dermis of the patient.

SUMMARY:
Mono-centre, open label (unblinded). 8 patients + 2 potential replacements. Duration up to 9 weeks: up to 6 weeks screening (42 days), 2 weeks of treatment (14 days, depending on sensor functionality) and 1 week of follow up (7 days)

DETAILED DESCRIPTION:
This study is an investigational study, which will be conducted only at one site in Germany. The investigators, the patient and the sponsor will be unblinded.

As soon as the eligibility of the patient is confirmed the patient is enrolled. The screening results are valid up to 42 days. Within that time the first measurement visit including the insertion of the device should be performed. If the first measurement visit is delayed a re-screening has to be performed. Should the patient not pass the re-screening, the patient is considered as a screening failure and must be excluded.

The trial is structured into three phases, the screening/enrolment phase, the insertion/measurement phase and the follow-up phase.

Screening/Enrolment Phase: 6 weeks (42 days), 1 visit

Insertion/Measurement phase: Up to 2 weeks (14days), up to 6 measurement visits

Follow-up Phase: 1 week (7 days), 1 visit

ELIGIBILITY:
Inclusion Criteria:

* Body mass index within the range of 19-40 kg/m2, inclusive
* Diabetes type 1 and 2
* Females (if of childbearing potential) must agree to abstain from sexual intercourse or use reliable forms of contraception e.g. condom or diaphragm with spermicide or oral contraceptives to prevent pregnancy during the study
* Signed written Informed Consent

Exclusion Criteria:

* Inability to follow the protocol schedule
* Participating in another clinical trial, if it is not a "non-investigational clinical study (NICS)
* Pregnant or lactating females,
* Any known hypersensitivity to any of the products used in the study, including preservatives etc.
* Malignancies requiring therapy during the study
* Severe chronic diseases e.g. renal failure, liver cirrhosis etc. which may interfere with the conduct or completion of the study
* Acute severe infection disease at the time of enrolment
* Alcohol and/or drug abuses
* Vulnerable patients (e.g. persons kept in detention)
* Poorly controlled diabetes mellitus with hemoglobin A1C higher than 10%

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Correlation between blood glucose and interstitial fluid (ISF) glucose concentration | 6 measurements within 14 days
  Mean absolute relative difference (MARD) of fluorescence sensor values and laboratory blood glucose values
Adverse event reporting | 14 days
  Incidence of reported ADE, with focus on number of SADE

SECONDARY OUTCOMES:
Lag time | 6 measurements within 14 days
  Determine changes in blood glucose to fluorescence lag time (in minutes)
Stability of measurements | 6 measurements within 14 days
  Stability of the FiberSense fluorescence measurement signals over the wearing time
Correlation between the fluorescence readings of the sensor and capillary blood glucose measurements | 6 measurements within 14 days
  Mean absolute relative difference (MARD) of fluorescence sensor values and capillary blood glucose values
Signal to noise ratio | 6 measurements within 14 days
Signal drift | 6 measurements within 14 days
Patient impression | after 14 days
  Subjective impression of the patients assesed by 5/6-point scale

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hasslacher, Prof. Dr., Principal Investigator — Diabetesinstitut Heidelberg
Locations (1):
- Diabetes Instiut Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No